CLINICAL TRIAL: NCT04366687
Title: Smart Parents--Safe and Healthy Kids: Small RCT
Brief Title: Smart Parents--Safe and Healthy Kids
Acronym: SPSHK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Penn State University (Other)
Responsible Party: Principal Investigator, Katelyn Guastaferro, Assistant Research Professor, Penn State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CMSN 8875
Record Dates: First submitted 2020-04-09; First posted 2020-04-29 (Actual); Last update posted 2020-04-29 (Actual); Status verified 2020-04

CONDITIONS: Child Sexual Abuse
Keywords: child sexual abuse; prevention; parenting; intervention science

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PAT-AU (Active Comparator): Parents randomized to this arm (i.e., group) receive Parents as Teachers (PAT) services as usual (AU).
  Interventions: Behavioral: Parents as Teachers
- PAT+CSA (Experimental): Parents randomized to this arm (i.e., group) receive the added CSA-focused session (Smart Parents - Safe and Healthy Kids) added to typical Parents as Teachers (PAT).
  Interventions: Behavioral: Smart Parents - Safe and Healthy Kids

INTERVENTIONS:
Behavioral: Smart Parents - Safe and Healthy Kids — Smart Parents - Safe and Healthy Kids (SPHSK) is a module designed to be added to existing evidence-based parent education programs. Because the module builds off of the core parenting skills developed in existing parent education programs, the module can be delivered in one session. SPSHK is comprised of three key CSA-prevention components: healthy child sexual development, parent-child communication about sex and sexual behaviors, and CSA-specific safety strategies such as vetting a babysitter and monitoring one-on-one time with adults. Behaviorally based, the module presents developmentally comprehensive information to parents of children 0-13 and utilizes role-playing scenarios and activities to maximize parents' use of learned skills.
  Arms: PAT+CSA
Behavioral: Parents as Teachers — Parents as Teachers (PAT) is a parent-support program delivered to parents of children under five and focuses on improving parenting skills through parent-child interactions, development centered parenting, and general well-being. PAT has demonstrated positive effects on child and parent outcomes related to school readiness.
  Arms: PAT-AU

SUMMARY:
The purpose of the proposed study is to assess the effectiveness of the addition of a single-session child sexual abuse (CSA) prevention module (Smart Parents - Safe and Healthy Kids) on improving parents' knowledge, attitudes, and behaviors regarding CSA prevention for parents already receiving parent-education services. The investigators hypothesize that parents who receive the parenting curriculum and the CSA prevention module will (a) demonstrate significant improvement in CSA-related awareness (i.e., knowledge, attitudes) and protective behaviors from pre-test to post-test, and (b) demonstrate higher scores on CSA-related awareness and protective behaviors as compared to parents who only receive the parenting curriculum.

ELIGIBILITY:
Inclusion Criteria:

1. Parent or caregiver > 18 years old
2. Parent or caregiver of at least one child under 13
3. Enrolled in PAT

Exclusion Criteria:

1. Parent/caregiver does not speak English
2. Parent is mandated (i.e., court-ordered) to attend parent-training program

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2018-04-02 (Actual); Primary Completion 2019-11-08 (Actual); Study Completion 2019-11-08 (Actual)

PRIMARY OUTCOMES:
Change in SmartParents' Knowledge (ASK): Awareness Factor | through study completion, an average of 14 weeks
  This factor measures change in parents' self-reported knowledge of CSA and positive attitudes toward CSA prevention, operationally defined henceforth as 'awareness'
Change in SmartParents' Knowledge (ASK): Protective Behaviors Factor | through study completion, an average of 14 weeks
  This factor measures change in parents' self-reported use of protective behaviors to limit risk for CSA.

SECONDARY OUTCOMES:
Change in Alabama Parenting Questionnaire: Involvement | through study completion, an average of 14 weeks
  e.g., "You ask your child about his/her day in school"
Change in Alabama Parenting Questionnaire: Positive Parenting | through study completion, an average of 14 weeks
  e.g., "You hug or kiss your child when he/she does something well"
Change in Alabama Parenting Questionnaire: Inconsistent Discipline | through study completion, an average of 14 weeks
  e.g., "The punishment you give your child depends on your mood"

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Guidance Resource Center Bradford, Bradford, Pennsylvania
  - Guidance Resource Center DuBois, DuBois, Pennsylvania
  - Wesley Family Services, Greensburg, Pennsylvania
  - Greater Nanticoke Area Family Center, Nanticoke, Pennsylvania
  - Youth Service Bureau, State College, Pennsylvania
  - Greater Susquehanna Valley United Way, Sunbury, Pennsylvania

REFERENCES:
- [Background] Guastaferro K, Zadzora KM, Reader JM, Shanley J, Noll JG. A Parent-focused Child Sexual Abuse Prevention Program: Development, Acceptability, and Feasibility. J Child Fam Stud. 2019 Jul;28(7):1862-1877. doi: 10.1007/s10826-019-01410-y. Epub 2019 Apr 18. PMID 31662600

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-01-15): https://cdn.clinicaltrials.gov/large-docs/87/NCT04366687/Prot_SAP_000.pdf
  • Informed Consent Form (2019-01-15): https://cdn.clinicaltrials.gov/large-docs/87/NCT04366687/ICF_001.pdf